CLINICAL TRIAL: NCT07257835
Title: Dupilumab Therapy for Refractory Eosinophilic Gastrointestinal Disorders in Children
Brief Title: Dupilumab Therapy for EGIDs
Status: Recruiting | Type: Observational
Sponsor: Children's Hospital of Fudan University (Other)
Responsible Party: Principal Investigator, Ying HUANG, Head of gastroenterology department, Children's Hospital of Fudan University
Other Study IDs: Dupilumab in EGIDs
Record Dates: First submitted 2025-08-21; First posted 2025-12-02 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: Eosinophilic Gastrointestinal Disorders (EGIDs)
MeSH Terms: conditions — Eosinophilic Esophagitis | interventions — dupilumab; Injections, Subcutaneous

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — blood sample, stool samples and biopsy samples during endoscopy
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: Yes

GROUPS / COHORTS (1):
- The patient is over 1 year old; for those who do not respond to conventional treatments (proton pump
  Interventions: Drug: Dupilumab - Standard Dose; Device: subcutaneous injection

INTERVENTIONS:
Drug: Dupilumab - Standard Dose — Dose: For patients with weight ≥ 15kg but < 30kg, take 200mg each time, every two weeks; for those with weight ≤ 30kg but < 60kg, take 300mg each time, every two weeks; for those with weight ≥ 60kg, take 300mg each time, once a week.
Device: subcutaneous injection — Dose: For patients with weight ≥ 15kg but < 30kg, take 200mg each time, every two weeks; for those with weight ≤ 30kg but < 60kg, take 300mg each time, every two weeks; for those with weight ≥ 60kg, take 300mg each time, once a week.

SUMMARY:
This is a single-center observational study to investigate the efficacy and tolerability of dupilumab in children with refractory eosinophilic gastrointestinal disorders.

DETAILED DESCRIPTION:
Eosinophilic Gastrointestinal Disorders (EGIDs) are chronic inflammatory diseases caused by extensive infiltration of eosinophils in the gastrointestinal tract. Treatment requires long-term dietary avoidance, long-term oral administration of high-dose omeprazole, as well as hormones and immunosuppressants, but the results are unsatisfactory and the side effects are significant. Dupilumab is a fully human monoclonal antibody (IgG4 type) that can specifically bind to the IL-4Rα subunit shared by the IL-4 and IL-13 receptor complexes to inhibit the signal transduction of IL-4 and IL-13. Current studies have shown that subcutaneous treatment with dupilumab for eosinophilic esophagitis has significant efficacy. In recent years, this drug has been reported to be used for various forms of gastrointestinal diseases such as eosinophilic gastritis, duodenitis, etc., with remarkable efficacy. In recent years, there has been an increasing number of children with refractory eosinophilic gastrointestinal diseases, which can easily cause repeated large ulcers, perforation, and stenosis in the gastrointestinal tract, requiring surgical intervention. This disease seriously affects the growth and development of children and urgently requires better treatment options. This study aims to evaluate the efficacy and tolerance of dupilumab in children with refractory eosinophilic gastrointestinal diseases.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of Refractory Peptic Ulcers
* with Refractory Eosinophilic Gastrointestinal Disorders

Exclusion Criteria:

* with Active Helicobacter pylori infection at present.
* with Inflammatory bowel disease
* with Parasite infection
* with Cancer

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children diagnosed with refractory eosinophilic gastrointestinal disorders who were seen at the Children's hospital of Fudan university who met the inclusion and exclusion criteria would be enrolled in this study.
Sampling Method: Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2025-01-01 (Actual); Primary Completion 2027-01-01 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
Endoscopic response rate | week12, week26, week52
  The ulcer reaches stage S (healed) or stage H (healing period), or the ulcer area has decreased by more than 50%.

SECONDARY OUTCOMES:
Relative Change of Peak Eosinophil Counts in the Stomach | week12，week26，week52
  We will determine the relative change from baseline in the peak eosinophil count in the five high-power fields (HPFs) with the highest eosinophil density in the antrum and/or body of the stomach after intervention.

OTHER OUTCOMES:
Adverse event | within one year
  The rate of the potential adverse events were monitored during the intervention.

CONTACTS AND LOCATIONS:
Locations (1):
- 201102, Shanghai, China

IPD SHARING:
Plan to Share IPD: Undecided